CLINICAL TRIAL: NCT01739569
Title: Long-term Effect of Healthy Lunch and Snack Meal on Reaction Time and Well-being: A Randomised Controlled Intervention in Physicians and Nursing Staff.
Brief Title: Effect of Healthy Lunch and Snack Meal on Reaction Time and Well-being of Physicians and Nursing Staff (Go-No-Go)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Christian Bitz, Head of Research, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: EFFECT.A01.2012
Record Dates: First submitted 2012-11-22; First posted 2012-12-03 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Nutrition Intervention
Keywords: Diet treatment; Mental Health; Reaction time; State of moods; Working hours; Medical Hospital Staff
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary treatment (Experimental): Dietary treatment with healthy lunch and snack meal during working hours
  Interventions: Other: Dietary treatment
- Habitual meals (No Intervention): Dietary treatment with habitual diet

INTERVENTIONS:
Other: Dietary treatment — Dietary treatment with healthy lunch and snack meal during working hours
  Arms: Dietary treatment

SUMMARY:
The aim of this study is to investigate the impact of increased availability of healthy food and drink during working hours on reaction time and well-being in physicians and nursing staff.

Hospital medical staff often works long and hectic hours, without adequate meal or rest breaks in order to provide 24-hour care. This is a concern, as not only the staff's well-being is important to the individual welfare, but it is also vital to the quality and safety of the care their patients receive. The investigators believe that by focusing on physicians and nursing staffs nutrition the investigators will see a positive effect on staff performance and well-being - and thus ultimately possibly on patient safety.

Hypothesis: The provision of healthy lunch and snack meal during working hours for a period of 4 weeks will improve reaction time and well-being compared to habitual diet in physicians, nurses and nursing assistants.

DETAILED DESCRIPTION:
The study is designed as a randomised controlled 2 x 4 weeks cross-over trial, initiated with a 1-week run-in period. The study sample will consist of 60 volunteer physicians, nurses and nursing assistants from Herlev University Hospital in Copenhagen, Denmark. A healthy lunch and snack meal meeting the current danish diet recommendations will be delivered daily during all working days in the intervention period. During the control period, the participants are requested to maintain their habitual dietary intake at work. Reaction time will be assessed by reaction time test Go/No-Go, a subtest of Test-battery for Attention Performance. Changes in mood will be measured by the Profile of Mood State questionnaire. In addition, dietary intake, level of physical activity and palatability of the intervention diet will be registered.

ELIGIBILITY:
Inclusion Criteria:

* Employed in Herlev University Hospital as physician, nurse or nursing assistant (males and females)
* Age 20-70 years
* BMI 18,5-30 kg/m2
* Work at least 30 h/wk
* Have daily contact with patients and/or have responsibilities that may affect patient safety
* Primarily work in day- or evening shifts during the study period
* Not having any intentions of loosing weight or changing lifestyle habits during the study period
* Not suffer from any diseases that might affect dietary intake (e.g. food allergies, food intolerance)
* Not dine in the staff canteen, the Diastole, more than once a week
* Be able to write and understand the Danish language

Exclusion Criteria:

* For those working >35 h/wk having holiday/ time off duty for more than 9 consecutive days during the study period.
* For those working <35 h/wk having holiday/time off duty for more than 5 consecutive days during the study period
* Not to be able to attend the planned tests in the study
* Pregnancy
* Intensive physical exercise (e.g. strength training) > 5 hours/wk
* Suffer from food allergies or - intolerance

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Reaction-time | week 0, week 5 and week 9
  Differences in reaction-time, as measured by the reaction time test Go/No-Go, a subtest of Test-battery for Attentional Performance from baseline (week 0) to week 4 in the intervention period and week 4 in the control period.

SECONDARY OUTCOMES:
Dietary intake | Week 0, week 5, week 9
  Differences in dietary intake with respect to macronutrient composition, meal pattern and choice of food items measured by self-reported records during 4 working days using a standardized dietary record form
Physical activity | Week 0, week 5, week 9
  Differences in 24-hours physical activity measured by self-reported records during four working days using a standardized physical activity record form.
Palatability of the diet eaten during working hours | Week 0, week 5 and week 9
  Differences in palatability of the intervention diet compared to the control diet measured by scores using a specific and standardized Visual Analouge Scale (VAS-scores).
Well-being | Week 0, week 5 and week 9
  Differences in selfreported well-being, as measured by the POMS Questionaire (McNair et.al. Manual of the Profile of Mood States. San Diego:Educational and Industrial Testing Service;1981) form baseline (week 0) to week 4 in the intervention period and week 4 in the control period.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Bitz, Cand Scient, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- EFFECT, Copenhagen University Hospital at Herlev, Herlev, Copenhagen, Denmark

REFERENCES:
- [Result] Leedo E, Beck AM, Astrup A, Lassen AD. The effectiveness of healthy meals at work on reaction time, mood and dietary intake: a randomised cross-over study in daytime and shift workers at an university hospital. Br J Nutr. 2017 Jul;118(2):121-129. doi: 10.1017/S000711451700191X. PMID 28820084